CLINICAL TRIAL: NCT06759597
Title: Macular Changes After Phacoemulsification in Patients with Neovascular AMD
Brief Title: The Effect of Phacoemulsification on the Macular Changes in Patients with Neovascular Age-related Macular Degeneration
Acronym: it does not
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Demiana alkes zakka labib, doctor, Assiut University
Other Study IDs: Macular Changes after PHE
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Neovascular (wet) Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The macula has a very high concentration of photoreceptor cells - the cells that detect light. They send signals to the brain, which interprets them as images. The rest of the retina processes our peripheral, or side vision To explore whether cataract surgery evokes development or relapse of choroidal neovascularization (CNV) in wet age-related macular degeneration (AMD) patients followed for a 1-year postoperative period

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) is a leading cause of vision loss in adults over the age of 50. AMD causes damage to a small part of the retina responsible for central vision called the macula. When damage to the macula occurs, it typically causes loss of central, detailed vision which results in difficulty with tasks such as reading, driving, threading a needle, or recognizing faces.

Phacoemulsification is a modern-day cataract surgery that employs ultrasound energy to emulsify the nucleus, vacuum to catch the nuclear material, and irrigation and aspiration for cortex and viscoelastic removal.

It is currently impossible to draw definitive conclusions whether phacoemulsification (PhE) is safe for people with age-related macular degeneration (ARMD). It is not clear if PhE causes the progression of ARMD and affects visual acuity (VA). The purpose was to analyze the possible association of PhE with ARMD progression in the early and late (up to 18 months after surgery) period.

ELIGIBILITY:
Inclusion Criteria:Subjects included in this study aged above 50 and presented for routine check up after undergoing phacoemulsification:

* Above 50 years old

  * not diabetic individuals
  * wet ARMD

Exclusion Criteria:

* intraoperative complications

  * Eyes with diseases predisposing them for postoperative macular edema, preexisting macular edema, and eyes that developed cystoid macular edema
  * active ocular inflammation or infection _glaucoma
  * A preoperatively worsened VA regardless phE
  * ocular trauma
  * patients with central retinal ischemia
  * previous vitrectomy
  * dry amd

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: old age population had phacoemulsefcation with history of neovascular AMD
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
To figure out the possibility of Postoperative conversion or relapse ( Dry to wet , wet to reactivated CNV) | baseline
  To explore whether cataract surgery evokes development or relapse of choroidal neovascularization (CNV) in wet age-related macular degeneration (AMD) patients followed for a 1-year postoperative period

REFERENCES:
- See also: Related Info — https://scholar.google.com.eg/scholar?q=CATARACT+SURGERY+AND+NEOVASCULAR+AGE-RELATED+MACULAR+DEGENERATION+DEVELOPMENT+OR+EXACERBATION:+A+RETROSPECTIVE+ANALYSIS&hl=en&as_sdt=0&as_vis=1&oi=scholart#d=gs_qabs&t=1735601011755&u=%23p%3DcqNfzWRFpsEJ